CLINICAL TRIAL: NCT06723704
Title: Prognosis in Adult Patients with Congenital Heart Disease: an Observational Study
Brief Title: Prognosis in Adult Patients with Congenital Heart Disease
Acronym: PRO-ACHD
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Graziani Francesca, MD, PhD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 4742
Record Dates: First submitted 2024-11-28; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Adult Congenital Heart Disease
Keywords: adult congenital heart disease; ACHD; prognosis; long-term; follow-up
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ACHD cohort: Adult patients with congenital heart disease either untreated, corrected or palliated, evaluated in our ACHD Outpatient Clinic between 2014 and 2026 with at least one-year follow-up.

SUMMARY:
This is a mono-center observational ambispective study in which adult patients with congenital heart disease evaluated at our institution will be enrolled.

The primary endopoint is to assess the clinical and echocardiographic predictors of adverse events during follow-up (death, arrhythmias, cardiac hospitalization).

The secondary endpoints are: 1) evaluation of the incidence of the singular components of the primary endpoint; 2) evaluation of the prognostic impact of acquired lesions, including valve disease not present at birth; 3) need for surgical/percutaneous interventions during follow up.

Participants will be evaluated in the context of scheduled follow-up visits in our Outpatient ACHD Clinic. No interventions/drug administration will be performed other than those required by standard clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients evaluated in our ACHD Outpatient Clinic between January 2014 and December 2026
* Age ≥ 18 years

Exclusion Criteria:

* Patients without congenital heart disease confirmed during the first evaluation
* Impossibility to retrieve information about the first clinical evaluation in our clinic from our electonic datasets
* Follow up shorter than one-year
* Refused consent to participate to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pazients with congenital heart disease either untreated, corrected or palliated evaluated for the first time in our ACHD Oupatient Clinic during the study period
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
cardiovascular outcomes | 5 years
  composite endpoint of death and cardiac hospitalization
major cardiac arrhytmias | 5 years
  occurence of ventricular and/or atrial arrhythmias

SECONDARY OUTCOMES:
changes in echocardiographic parameters over time | 12 months
  * variations in cardiac chamber size (volumes in ml, diameters in mm);
  * variations in left ventricular function (assessed as left ventricular ejection fraction in % using the Simpson biplane method);
  * variations in right ventricular systolic function (assessed as tricuspid anular plane systolic excursion in mm).
heart valve disease (new-onset or progression) | 12 months
  progression of pre-existing heart valve disease or new-onset valve dysfunction assessed through echocardiography

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin YS, Liu PH, Wu LS, Chen YM, Chang CJ, Chu PH. Major adverse cardiovascular events in adult congenital heart disease: a population-based follow-up study from Taiwan. BMC Cardiovasc Disord. 2014 Mar 21;14:38. doi: 10.1186/1471-2261-14-38. PMID 24655794
- [Background] Diller GP, Kempny A, Alonso-Gonzalez R, Swan L, Uebing A, Li W, Babu-Narayan S, Wort SJ, Dimopoulos K, Gatzoulis MA. Survival Prospects and Circumstances of Death in Contemporary Adult Congenital Heart Disease Patients Under Follow-Up at a Large Tertiary Centre. Circulation. 2015 Dec 1;132(22):2118-25. doi: 10.1161/CIRCULATIONAHA.115.017202. Epub 2015 Sep 14. PMID 26369353
- [Background] Lytzen R, Vejlstrup N, Bjerre J, Petersen OB, Leenskjold S, Dodd JK, Jorgensen FS, Sondergaard L. Live-Born Major Congenital Heart Disease in Denmark: Incidence, Detection Rate, and Termination of Pregnancy Rate From 1996 to 2013. JAMA Cardiol. 2018 Sep 1;3(9):829-837. doi: 10.1001/jamacardio.2018.2009. PMID 30027209
- [Background] van der Linde D, Konings EE, Slager MA, Witsenburg M, Helbing WA, Takkenberg JJ, Roos-Hesselink JW. Birth prevalence of congenital heart disease worldwide: a systematic review and meta-analysis. J Am Coll Cardiol. 2011 Nov 15;58(21):2241-7. doi: 10.1016/j.jacc.2011.08.025. PMID 22078432
- [Background] Warnes CA, Liberthson R, Danielson GK, Dore A, Harris L, Hoffman JI, Somerville J, Williams RG, Webb GD. Task force 1: the changing profile of congenital heart disease in adult life. J Am Coll Cardiol. 2001 Apr;37(5):1170-5. doi: 10.1016/s0735-1097(01)01272-4. No abstract available. PMID 11300418
- [Background] Moons P, Bovijn L, Budts W, Belmans A, Gewillig M. Temporal trends in survival to adulthood among patients born with congenital heart disease from 1970 to 1992 in Belgium. Circulation. 2010 Nov 30;122(22):2264-72. doi: 10.1161/CIRCULATIONAHA.110.946343. Epub 2010 Nov 22. PMID 21098444